CLINICAL TRIAL: NCT03251586
Title: Test-Retest Reliability of oVEMP's Across Different Electrode Montages
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to time constraints, the study will not be able to be completed as outlined
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Makowiec, Vestibular Fellow, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140805
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Vestibular Abnormality; Vestibular Nerve Disorders
MeSH Terms: conditions — Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (8):
- 20-29 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 30-39 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 40-49 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 50-59 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 60-69 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 70-79 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 80-89 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage
- 90-99 (Experimental): Participants within the above age range who have normal hearing and no history of balance disorders or unsteadiness.
  Interventions: Diagnostic Test: oVEMP - infra-orbital electrode montage; Diagnostic Test: oVEMP - belly-tendon electrode montage

INTERVENTIONS:
Diagnostic Test: oVEMP - infra-orbital electrode montage — oVEMPs are short latency (~10 ms) stimulus-synchronized extra-ocular muscle reflexes produced in response to appropriate stimuli. The response is believed to originate from excitation of the utricular macula with the subsequent neural response relayed to the brain by the superior portion of the vestibular nerve. Changes in the electrical field of the contralateral inferior oblique muscle can be recorded by an electrode placed at the infra-ocular midline of the lower lid while having the subject gaze upward. The conventional electrode montage, the infra-orbital electrode montage, has the active electrode placed directly inferior to the eye and the reference electrode placed 2-3 cm below the active on the cheek. This electrode montage may result in reference contamination, which will cause an artificially reduced amplitude response, as a portion of the response can be measured by the reference electrode.
Diagnostic Test: oVEMP - belly-tendon electrode montage — oVEMPs are short latency (~10 ms) stimulus-synchronized extra-ocular muscle reflexes produced in response to appropriate stimuli. The response is believed to originate from excitation of the utricular macula with the subsequent neural response relayed to the brain by the superior portion of the vestibular nerve. Changes in the electrical field of the contralateral inferior oblique muscle can be recorded by an electrode placed at the infra-ocular midline of the lower lid while having the subject gaze upward. The belly-tendon electrode montage consists of an active electrode placed laterally to the midline of the lower eyelid and a reference electrode placed on the inner canthus. This reference location is believed to be electrically neutral, and should therefore result in larger amplitude responses as the response would not be subject to reference contamination.

SUMMARY:
"Test-Retest Reliability of ocular vestibular evoked myogenic potentials (oVEMPs) across different electrode montages."

The purpose of this project is to compare the response characteristics of the ocular vestibular evoked myogenic potential in patients grouped by decade (i.e. 20's-90's) using two different recording montages and two different stimulus types (i.e. air and bone conducted sound). The long-term goal is to increase the sensitivity and specificity of the oVEMP when used clinically to identify vestibular disorders affecting the utricle and superior portion of the vestibular nerve.

.

DETAILED DESCRIPTION:
Specific Aim: Compare the difference in the contralateral peak-to-peak N1-P1 amplitude and N1 latency between the belly tendon electrode montage with the conventional infraorbital electrode montage in otologically normal patients grouped by decade with the goal of developing normative values to use clinically.

The oVEMP is a short latency (~10 ms), negative polarity evoked myogenic potential that is recorded from the extraocular muscles. The oVEMP test is well-tolerated by patients and is simple to administer. Whereas the recording of the cVEMP to air-conducted stimuli represents a means for evaluating the function of the saccule and inferior vestibular nerve, the oVEMP in response to mechanical, and probably air conducted stimuli, is now felt to represent a method for assessing the functional integrity of the utricle and superior vestibular nerve.

The oVEMP response is recorded from beneath both the ipsilateral and contralateral eyes, but the largest response is typically seen in the contralateral recording. The contralateral utricular-ocular pathway terminates on the inferior oblique muscle, the electrical field of which can be recorded by an electrode placed at the midline of the lower lid and having the subject gaze upward (i.e. which results in the inferior oblique muscle becoming more superficial to the location of the surface electrode.

The the absolute oVEMP N1 peak-to-peak amplitude has become the most important measurement for diagnostic purposes. Typical oVEMP latencies are ~11 ms for the negative peak (N1) and ~15 ms for the following positive peak (P1) .

Variables that may confound recording oVEMPs include body position and electrode montages. Regarding electrode placement, there are three different electrode montages that have been studied and implemented clinically. The vast majority of clinics favor the electrode montage reported in the early papers describing the oVEMP. The authors reported that the non-inverting electrode was placed infraorbitally at the margin of the lower eyelid. The inverting electrode was placed 2 cm inferior to the location of the non-inverting electrode. Two additional electrode montages that have been reported include: 1) the noninverting electrodes placed at the margin of the lower eyelid slightly lateral to midline and the inverting electrode placed rostral to the inner canthus of the eye, and, 2) the noninverting electrodes placed at the middle of the lmargin of the lower eyelid and a single common inverting electrode placed on the chin. A report by Sandhu et al. (2013) indicated that the maximal oVEMP amplitude was recorded with the former electrode montage. In this montage, the inverting electrode is placed over a tendon, which is believed to be (relatively) electrically neutral.

Skin surface electrodes are sensitive to the desired muscle activity (i.e. signal) recorded locally as well as non-stimulus-related electrical activity (i.e. noise) that can be both endogenous and exogenous. Where the signal is common to both the inverting and non-inverting electrodes this activity routed into a differential electrode can result in cancellation of some or all of the desired signal.

Recently published data from our laboratory has shown that the Sandhu montage (i.e. the "belly-tendon electrode montage) in the sitting position is the optimal method for testing patients who are otologically and neurologically normal. This montage is associated with a larger N1 amplitude and a larger peak-to-peak amplitude for oVEMP measurements for young, normal patients. Due to the knowledge that the amplitude of the oVEMP response decreases with age, however, normative values based on decade would be necessary to have the oVEMP response be as clinically useful as possible.

Significance and Potential of the Research:

Establishing normative values based on decade will allow for higher sensitivity and specificity to vestibular impairments affecting the utricle and superior portion of the vestibular nerve, as well as increase the sensitivity and specificity to disorders such as Superior Semicircular Canal Dehiscence Syndrome.

Methods:

Subjects: Participants will include groups of patients between 20-90 years of age. The groups will be composed of 10-15 subjects per group to allow for normative data to be calculated. Participants will be recruited by phone using databases housed in the Odess Otolaryngology Department at Vanderbilt Bill Wilkerson Center, via flyers posted at Vanderbilt University Medical Center, and through Research Match email blasts. The study protocol will undergo review by the Vanderbilt Institutional Review Board (submitted-see Appendix).

oVEMP Recording: For the oVEMP recording (utricular assessment), subjects will be seated in a comfortable reclining will be compared during this study. First, an electrode montage and recording parameters similar to those reported by Chihara et al. (2007) will be used to record the oVEMP. Disposable silver/silverchloride electrodes will be placed infraorbitally beneath each eye (i.e., infraorbital 1 cm) representing the non-inverting amplifier inputs and 3cm infraorbitally will serve as the location for the inverting electrode. A second electrode montage with recording parameters similar those reported by Sandhu et al. (2013) will be used simultaneously to record oVEMP responses. Disposable silver/silverchloride electrodes will be placed on the belly of the inferior oblique muscle representing the non-inverting amplifier inputs and the tendon of the inferior oblique muscle will serve as the location for the inverting electrode. The ground electrode will be placed at Fpz for both electrode montages.

When recording the oVEMP, the subjects will be seated and instructed to keep their head at midline and gaze at a target positioned ~30° upward at midline. During the recording, the investigator will monitor to ensure the subject's chin is parallel to the horizon. Stimuli for the oVEMP recordings will be presented monaurally through Etymotic ER-3A insert earphones or a B81 bone conductor and consist of 500 Hz tone bursts presented at a rate of 5.1/sec. The tone burst will have a 2 cycle rise time, 1 cycle plateau and a 2 cycle fall time. A Neuroscan (Herndon, UA) multi-channel evoked potential recording system will enable us to record simultaneously the oVEMP response from each of the two electrode montages. EMG activity will be amplified by 100,000 times and signal averaged over 100 msec. A minimum of 120 individual samples will be collected for each recording. Each tracing will be replicated at least one time so that the waveform reproducibility can be estimated. Order effects will be eliminated by counterbalancing the order of the starting ear. oVEMPs from the two electrode montages will be recorded simultaneously, so counterbalancing the electrode montage will be unnecessary. A minimum of two amplitude measures will be completed for each electrode montage condition in each position, for a total minimum of 8 recordings per subject. The subject will be given 1-2 minutes to rest their eyes between recordings.

Stimulus level will be calibrated in dBpeak SPL using a 2-cm3 coupler to a sound-level meter (Bruel & Kjaer). The stimulus waveforms and amplitude spectra will be measured by routing the air conduction output of the sound-level meter to a spectrum analyzer.

Statistical Methods:

Analysis: Summary statistics will be provided for all demographic and clinical variables, along with 95% confidence intervals and side-by-side boxplots. Between-group differences in categorical variables will be assessed via chi-squared tests while differences in continuous variables will be assessed via the Wilcoxin rank-sum test (using significance level alpha = 0.0125 in primary analysis as per the power calculation above). Hotelling's T-squared distribution will also be used as an omnibus or simultaneous test that the groups are the same for all variables in the primary analysis. Amplitude differences obtained using each montage will be calculated as a change expressed in percentage using the formula below:

(n1-p1 amplitude montage2 - n1-p1 amplitude montage 1)

--------------------------------------------------------------- n1-p1 amplitude montage 1

All statistical analyses will be performed with SPSS 23.

Facilities Available: The Vanderbilt Balance Disorders Laboratory is located in the Bill Wilkerson Center. The Balance Disorders Laboratory is equipped with state-of-the art equipment for comprehensive assessment of vestibular and auditory disorders. The facility includes a sound treated room, five diagnostic audiometers, five compact disk players for speech audiometry, five immittance meters, three otoacoustic emissions devices, two rotary vestibular test chairs, three videonystagmography systems, a computerized electronystagmography system, a computerized dynamic posturography system, a Neuroscan evoked response system with capability for 64 channel simultaneous brain signal acquisition, and 4 2-channel clinical evoked potentials systems.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing and no history of balance disorders

Exclusion Criteria:

* Hearing loss, a large amount of ear wax, inner ear of balance problems, and/or no recordable eye muscle responses

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Development of Normative Values per Decade | 5 months for data collection, one visit per subject.
  The oVEMP N1-P1 amplitude and N1 latency will be measured for each subject and will be used to calculate normative values for each decade. The goal is to provide clinics with normative information to base clinical evaluations on.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn F Makowiec, AuD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Result] Chang CM, Cheng PW, Wang SJ, Young YH. Effects of repetition rate of bone-conducted vibration on ocular and cervical vestibular-evoked myogenic potentials. Clin Neurophysiol. 2010 Dec;121(12):2121-7. doi: 10.1016/j.clinph.2010.05.013. Epub 2010 Jun 11. PMID 20541460
- [Result] Chihara Y, Iwasaki S, Ushio M, Murofushi T. Vestibular-evoked extraocular potentials by air-conducted sound: another clinical test for vestibular function. Clin Neurophysiol. 2007 Dec;118(12):2745-51. doi: 10.1016/j.clinph.2007.08.005. Epub 2007 Oct 1. PMID 17905655
- [Result] Curthoys IS, Iwasaki S, Chihara Y, Ushio M, McGarvie LA, Burgess AM. The ocular vestibular-evoked myogenic potential to air-conducted sound; probable superior vestibular nerve origin. Clin Neurophysiol. 2011 Mar;122(3):611-616. doi: 10.1016/j.clinph.2010.07.018. Epub 2010 Aug 14. PMID 20709596
- [Result] Govender S, Rosengren SM, Colebatch JG. The effect of gaze direction on the ocular vestibular evoked myogenic potential produced by air-conducted sound. Clin Neurophysiol. 2009 Jul;120(7):1386-91. doi: 10.1016/j.clinph.2009.04.017. Epub 2009 May 22. PMID 19464947
- [Result] Makowiec K, McCaslin DL, Jacobson GP, Hatton K, Lee J. Effect of Electrode Montage and Head Position on Air-Conducted Ocular Vestibular Evoked Myogenic Potential. Am J Audiol. 2017 Jun 13;26(2):180-188. doi: 10.1044/2017_AJA-16-0108. PMID 28520834
- [Result] Kantner C, Gurkov R. Characteristics and clinical applications of ocular vestibular evoked myogenic potentials. Hear Res. 2012 Dec;294(1-2):55-63. doi: 10.1016/j.heares.2012.10.008. Epub 2012 Oct 30. PMID 23123220
- [Result] Murnane OD, Akin FW, Kelly KJ, Byrd S. Effects of stimulus and recording parameters on the air conduction ocular vestibular evoked myogenic potential. J Am Acad Audiol. 2011 Jul-Aug;22(7):469-80. doi: 10.3766/jaaa.22.7.7. PMID 21993052
- [Result] Nguyen KD, Welgampola MS, Carey JP. Test-retest reliability and age-related characteristics of the ocular and cervical vestibular evoked myogenic potential tests. Otol Neurotol. 2010 Jul;31(5):793-802. doi: 10.1097/MAO.0b013e3181e3d60e. PMID 20517167
- [Result] Piker EG, Jacobson GP, McCaslin DL, Hood LJ. Normal characteristics of the ocular vestibular evoked myogenic potential. J Am Acad Audiol. 2011 Apr;22(4):222-30. doi: 10.3766/jaaa.22.4.5. PMID 21586257
- [Result] Piker EG, Jacobson GP, Burkard RF, McCaslin DL, Hood LJ. Effects of age on the tuning of the cVEMP and oVEMP. Ear Hear. 2013 Nov-Dec;34(6):e65-73. doi: 10.1097/AUD.0b013e31828fc9f2. PMID 23673615
- [Result] Rosengren SM, McAngus Todd NP, Colebatch JG. Vestibular-evoked extraocular potentials produced by stimulation with bone-conducted sound. Clin Neurophysiol. 2005 Aug;116(8):1938-48. doi: 10.1016/j.clinph.2005.03.019. PMID 15979939
- [Result] Sandhu JS, George SR, Rea PA. The effect of electrode positioning on the ocular vestibular evoked myogenic potential to air-conducted sound. Clin Neurophysiol. 2013 Jun;124(6):1232-6. doi: 10.1016/j.clinph.2012.11.019. Epub 2013 Jan 18. PMID 23333609
- [Result] Todd NP, Rosengren SM, Aw ST, Colebatch JG. Ocular vestibular evoked myogenic potentials (OVEMPs) produced by air- and bone-conducted sound. Clin Neurophysiol. 2007 Feb;118(2):381-90. doi: 10.1016/j.clinph.2006.09.025. Epub 2006 Dec 1. PMID 17141563
- [Result] Welgampola MS, Carey JP. Waiting for the evidence: VEMP testing and the ability to differentiate utricular versus saccular function. Otolaryngol Head Neck Surg. 2010 Aug;143(2):281-3. doi: 10.1016/j.otohns.2010.05.024. PMID 20647135